CLINICAL TRIAL: NCT06282900
Title: Pain and Screen Addiction: The Relationship Between the Number of Pain Areas and Screen Addiction and Various Screen Used in University Students: A Cross-Sectional Study
Brief Title: Pain and Screen Addiction in University Students
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1/15
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Student
Keywords: Musculoskeletal Pain; Screen Time; Physical Activity
MeSH Terms: conditions — Musculoskeletal Pain; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Other: University students — A cross-sectional study (Level IV evidence) will be conducted at the university (Acibadem University, Turkey). All students at the university will be invited to respond to a self-administered online survey. The survey will be prepared via Google Forms.

SUMMARY:
One of the most important factors why young people spend inactive time is the time they spend in front of the screen. Sedentary screen time refers to time spent using a screen-based device, such as a computer, television, smartphone, or tablet while being sedentary in any environment. The last decade has seen a disturbing increase in the amount of time young people spend in front of screens. Research shows that musculoskeletal disorders in the hand, wrist, arm, and neck occur at a high rate due to long-term and repetitive use of the smartphone, one of the electronic devices. People with musculoskeletal pain often complain of more than one area of pain.

The primary purpose of this study is to investigate the relationship between university students' use of various screen-based devices, the time they spend in front of the screen, and the number of painful areas they report on the body. Our secondary aim is to evaluate the relationship between pain, and screen time, and physical activity level.

DETAILED DESCRIPTION:
University is also an important year in individuals' lives because it is a period in which they gain autonomy and have more control over their own lives and behaviors. It is known that adult individuals have a decrease in their physical activity due to their work lives and responsibilities. For this reason, the increase in sedentary life has also become evident in early adulthood.

Sedentary living is associated with many health risks independent of physical activity, and physical activity directly affects health status. Since a large portion of the world's population is physically inactive, physical inactivity is considered a public health problem rather than an individual problem.

One of the most important factors why young people spend inactive time is the time they spend in front of the screen. Sedentary screen time refers to time spent using a screen-based device, such as a computer, television, smartphone, or tablet while being sedentary in any environment. The last decade has seen a disturbing increase in the amount of time young people spend in front of screens.

Most studies on screen addiction have focused on smartphone use. Smartphone addiction is positively associated with repetitive overuse of joints, leading to inflammatory changes in healthy joints. It can also affect proprioceptors in muscles and ligaments due to the postural problems it creates. Research shows that musculoskeletal disorders in the hand, wrist, arm, and neck occur at a high rate due to long-term and repetitive use of the smartphone, one of the electronic devices.

People who experience localized pain often report pain in other areas as well. Having pain in one area increases the risk of developing pain in other areas. Reporting more than one area of pain worsens the prognosis and increases the possibility of the current problem becoming chronic.

People with musculoskeletal pain often suffer from more than one site of pain, and compliance with standard definitions of widespread pain often excludes the majority with more than one site of pain.

The primary purpose of this study is to investigate the relationship between university students' use of various screen-based devices, the time they spend in front of the screen, and the number of painful areas they report on the body. Our secondary aim is to evaluate the relationship between pain and screen time, and physical activity level.

ELIGIBILITY:
Inclusion Criteria:

* All students between the ages of 18-25
* People who use screen-based devices for at least 2 hours a day

Exclusion Criteria:

* Presence of congenital deformity
* History of trauma to the musculoskeletal system in the last 6 months
* History of serious surgery
* Presence of neurological disease

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: All students between the ages of 18-25 who use screen-based devices for at least 2 hours a day will be included in the study. Those with congenital deformities, those who have experienced trauma to the musculoskeletal system in the last 6 months, and those with serious surgical or neurological diseases will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Investigating the use of screen-based devices | during the procedure
  Participants will be asked to rate the purpose of using screen-based devices (television, computer, game console, or hand-held electronic devices such as tablets and smartphones) during the day, how they use them, and their addictions on a 5-point Likert scale (0: strongly agree, 5: strongly disagree).
Musculoskeletal system evaluation | during the procedure
  The Extended Nordic Musculoskeletal Questionnaire will be used to record areas where participants experience pain due to static sitting posture issues such as prolonged sitting and screen use. The Extended Nordic Musculoskeletal Questionnaire consists of items related to nine body parts (neck, shoulders, upper back, elbows, wrists/hands, waist, hips/thighs, knees, ankles/feet) and includes questions about any time in the last 12 months, in the last 1 month, and during the day. Includes questions about experience. It evaluates upper body musculoskeletal symptoms associated with pain or numbness. The Extended Nordic Musculoskeletal Questionnaire generally uses a total score out of 100. High scores may indicate that ergonomic risks need to be evaluated and appropriate precautions taken.

SECONDARY OUTCOMES:
Physical activity assessment | during the procedure
  Participants' physical activity habits will be evaluated with the International Physical Activity Questionnaire (IPAQ - short form). The survey asks about activities that are done regularly at least once a week and how long it takes to do these activities. Activities recorded in the survey will be calculated in hour/week units and the intensity of the activities will be determined according to the MET (Metabolic Equivalent) values of the activities. Questionnaires will be scored using established methods published on the IPAQ website (www.ipaq.ki.se).
  The score obtained can help classify individuals into different activity levels:
  1. Low Level of Physical Activity: Total MET-minutes per week below 600.
  2. Moderate Level of Physical Activity: Total MET-minutes per week between 600 and 3000.
  3. High Level of Physical Activity: Total MET-minutes per week above 3000.

CONTACTS AND LOCATIONS:
Overall Officials: Elif E Safran, asst. prof., Study Director — Acibadem University
Locations (1):
- Acibadem University, Istanbul, None Selected, Turkey (Türkiye)